CLINICAL TRIAL: NCT06466304
Title: Inspiratory Muscle Training in Children With Beta Thalasemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Hagar Ahmed El-Hadidy, Physical Therapy for Internal Medicine and Geriatrics, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T -INT-06/2024- 544
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Beta Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): children patients with BTM accounted 20 children will receive two session per day of training by threshold inspiratory muscle trainer ( for six day per week for 12 weeks). the session will contain six sets of inspiratory muscle training and the one set will contain five respiratory cycles
  Interventions: Behavioral: inspiratory muscle training
- control group (No Intervention): children patients with BTM accounted 20 children will receive no trianiing and will serve as control children group

INTERVENTIONS:
Behavioral: inspiratory muscle training — children patients with BTM accounted 20 children will receive two session per day of training by threshold inspiratory muscle trainer ( for six day per week for 12 weeks). the session will contain six sets of inspiratory muscle training and the one set will contain five respiratory cycles
  Arms: study group

SUMMARY:
respiratory complications are very prevalent in children with beta thalasemia major (BTM), so choosing inspiratory muscle trianing to decrease of prevent it and to improve pulmoanry funntions is important

DETAILED DESCRIPTION:
children patients with BTM accounted 40 children will assigned to a group of inspiratory muscle training or waiting list group. the group will contain twenty children. the group of training will receive two session per day of training by threshold inspiratory muscle trainer ( for six day per week for 12 weeks)

ELIGIBILITY:
Inclusion Criteria:

* 40 beta thalassemia major children
* boys and girls

Exclusion Criteria:

* respiratory diseases
* cardiac diseases renal diseases liver diseases muscle and joint disease

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — self-representation of gender birth-certificate identity.
Enrollment: 40 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
forced expiratory volume t the first second of expiration | it will be assessed after 12 weeks
  it will measure pulmonary function

SECONDARY OUTCOMES:
forced vital capcity | it will be assessed after 12 weeks
  it will measure pulmonary function
FEV1/FVC | it will be assessed after 12 weeks
  it will measure pulmonary function
maximal inspiratory pressure | it will be assessed after 12 weeks
  it will measure strength of inspiratory muscles
six minute walk testing | it will be assessed after 12 weeks
  it will measure aerobic capacity
Pediatrics' Quality of Life Inventory (children proxy) | it will be assessed after 12 weeks
  it will assess quality of life and filled by children
Pediatrics' Quality of Life Inventory (parent proxy) | it will be assessed after 12 weeks
  it will assess quality of life and filled by parents of children

CONTACTS AND LOCATIONS:
Overall Officials: hagar el-hadidy, lecturer, Principal Investigator — Faculty of Physical Therapy, Ahram Canadian University (ACU), Giza, Egypt
Locations (1):
- Ahram canadian university, Giza, Egypt